CLINICAL TRIAL: NCT00550589
Title: Phase IIA Trial of 1% Topical Cidofovir for Treatment of High-Grade Perianal Squamous Intraepithelial Lesions in HIV-Infected Men and Women
Brief Title: Cidofovir in Treating HIV-Infected Patients With High-Grade Squamous Intraepithelial Lesions of the Skin Near the Anus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-046; U01CA121947 (NIH); CDR0000570720 (Other: NCI)
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Anal Cancer; Precancerous Condition
Keywords: high-grade squamous intraepithelial lesion; stage 0 anal cancer
MeSH Terms: conditions — Anus Neoplasms; Precancerous Conditions; Squamous Intraepithelial Lesions | interventions — Cidofovir; DNA Methylation; Gene Expression Profiling; Polymerase Chain Reaction; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir (Experimental): 1.0% topical cidofovir cream
  Interventions: Drug: cidofovir; Genetic: DNA methylation analysis; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Procedure: biopsy; Procedure: histopathologic examination

INTERVENTIONS:
Drug: cidofovir — 1.0% topical cream self-applied once daily for 5 consecutive days, with no treatment for the remaining 9 days (a treatment cycle). Subjects will receive up to 6 cycles of treatment.
Genetic: DNA methylation analysis — formalin fixed biopsy collected at baseline and 6 weeks after treatment discontinuation
Genetic: gene expression analysis — punch biopsy collected at baseline, after cycle 1, and 6 weeks after treatment discontinuation
Genetic: polymerase chain reaction — performed on punch biopsy specimens collected at baseline, after cycle 1, and 6 weeks after treatment discontinuation
Procedure: biopsy — punch biopsy collected at baseline, after cycle 1, and 6 weeks after treatment discontinuation
Procedure: histopathologic examination — Evaluated at baseline and 6 weeks after treatment discontinuation

SUMMARY:
RATIONALE: High-grade squamous intraepithelial lesions of the skin near the anus are caused by the human papillomavirus (HPV). Antiviral drugs,, such as cidofovir, act against viruses and may stop these lesions from becoming cancer.

PURPOSE: This phase II trial is studying the side effects and how well topical cidofovir works in treating HIV-infected patients with high-grade squamous intraepithelial lesions of the skin near the anus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the safety and tolerability of topical cidofovir in HIV-infected patients with perianal high-grade squamous intraepithelial lesions (HSIL).
* To estimate the regression rate of perianal HSIL in patients treated with this regimen.

Secondary

* To determine the human papilloma virus (HPV) DNA types and HPV strain variants present in perianal HSIL and normal perianal tissue.
* To determine if clinical regression of perianal HSIL is associated with clearance of HPV DNA.
* To identify the HPV DNA types present in the anus and cervix and compare them with the HPV DNA present in the perianus in order to determine if the HPV types associated with the perianal lesions are the same as those infecting the anus and cervix.
* To determine if there are abnormally methylated genes in perianal HSIL compared with normal perianal tissue and if these genes are the same or different from those that have been previously identified in anal and cervical dysplasia.
* To determine whether methylated genes are changed after treatment with cidofovir.
* To characterize differences in gene expression in perianal HSIL compared with normal perianal tissue.
* To examine changes in gene expression in perianal HSIL after exposure to cidofovir using RNA microarray analysis and confirm results with real-time polymerase chain reaction.
* To correlate pretreatment CD4 count, viral load, lesion size, methylation pattern, and/or HPV type and strain with the clinical efficacy of topical cidofovir.

OUTLINE: This is a multicenter study.

Patients apply topical cidofovir to the perianus once daily on days 1-5. Patients undergo punch biopsy of pretreatment lesional biopsy sites on day 14. Beginning 2-4 weeks after biopsy, patients receive course 2 of cidofovir therapy. Subsequent treatment repeats every 14 days for up to 6 courses* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive a total of 6 courses of study therapy.

Patients undergo collection of tumor and normal tissue for histopathological and molecular correlative studies. Punch biopsies are obtained at baseline, after the first course of therapy, and at 6 weeks after completion of therapy. Tissue samples are examined for histopathology, human papilloma virus (HPV)DNA typing, DNA methylation, and gene expression (via RNA microarray analysis and polymerase chain reaction).

After completion of study therapy, patients are followed at 6 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed perianal high-grade squamous intraepithelial lesions (HSIL) within the past 12 weeks

  * The perianal skin (i.e., perianus) is defined as extending radially 5 cm from the anal verge
  * Lesions must cover a surface area of ≥ 3 square centimeters
  * Lesions extending outside the perianus (e.g., vulvar lesions on the posterior perineum bordering the perianus) are allowed
* Serologic documentation of HIV infection AND meets 1 of the following criteria:

  * Has been on stable highly active anti-retroviral therapy (HAART) for ≥ 12 weeks prior to study entry
  * Has a CD4 count of > 200/mm³ AND is not receiving anti-retroviral therapy OR is currently receiving a non-HAART* anti-retroviral regimen with no plans to initiate HAART within the next 12 weeks NOTE: * A non-HAART regimen is considered to be a therapy that does not include a protease inhibitor or a non-nucleoside reverse transcriptase inhibitor
* No untreated invasive cancer of the lower genital tract
* No concurrent neoplasia requiring cytotoxic therapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 3 months
* Hemoglobin ≥ 8 g/dL
* ANC ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Creatinine < 1.5 times upper limit of normal (ULN)
* Total or conjugated (direct) bilirubin ≤ 2.5 times ULN
* AST and ALT ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No acute, opportunistic infection other than oral thrush, yeast vaginitis, or genital herpes within the past 14 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior ablative or surgical treatment of perianal dysplasia
* At least 4 weeks since prior topical treatment for perianal dysplasia

  * If any prior treatment caused significant trauma to ther area, healing should occur prior to starting treatment
* More than 14 days since prior acute treatment for infection (other than for oral thrush, yeast vaginitis, or genital herpes) or other serious medical illness
* No concurrent corticosteroids other than replacement doses
* No other concurrent investigational drugs except IND-approved anti-retroviral agents
* No concurrent systemic cytotoxic chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stier, MD, Study Chair — Boston Medical Center; Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Laser Surgery Care, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Result] Stier EA, Goldstone SE, Einstein MH, Jay N, Berry JM, Wilkin T, Lee JY, Darragh TM, Da Costa M, Panther L, Aboulafia D, Palefsky JM. Safety and efficacy of topical cidofovir to treat high-grade perianal and vulvar intraepithelial neoplasia in HIV-positive men and women. AIDS. 2013 Feb 20;27(4):545-51. doi: 10.1097/QAD.0b013e32835a9b16. PMID 23032420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cidofovir
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cidofovir
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Regression of Perianal High-grade Squamous Intraepithelial Lesions (HSIL)
Time Frame: 6 weeks after treatment discontinuation
Measure: Number; unit: proportion of participants
Arm/Group | Cidofovir
Number analyzed (Participants) | 33
proportion of participants | 0.515

2. Primary Outcome: Safety and Tolerability of Topical Cidofovir as Assessed by NCI CTCAE v3.0
Description: Number of study patients who had a serious adverse event
Time Frame: Every 2 weeks on study, 6 weeks after treatment discontinuation
Population: All enrolled patients
Measure: Number; unit: participants
Groups:
- Cidofovir: 1% cidofovir
Arm/Group | Cidofovir
Number analyzed (Participants) | 33
participants | 3

3. Secondary Outcome: Human Papilloma Virus (HPV) DNA Type in Perianal HSIL and Normal Perianal Tissue
Description: Number of patients with HPV16 at baseline in perianal HSIL and normal perianal tissue
Time Frame: Baseline
Population: Number of patients with tissue samples available at baseline
Measure: Number; unit: participants
Arm/Group | Cidofovir
Number analyzed (Participants) | 30
participants | 16

4. Secondary Outcome: Correlation of Clinical Regression of Perianal HSIL With Clearance of HPV DNA
Description: Number of patients who cleared HPV among those who had a complete or partial response
Time Frame: 6 weeks after treatment discontinuation
Population: Participants who had a partial or complete response and for whom pre and post-treatment HPV data were available
Measure: Number; unit: participants
Arm/Group | Cidofovir
Number analyzed (Participants) | 12
participants | 2

5. Secondary Outcome: Identification of HPV-DNA Types Present in the Anus
Description: Number of patients with HPV16 type present in the anus from anal swab or cytobrush at baseline
Time Frame: Baseline
Population: Number of patients with anal swabs or cytobrush results at baseline
Measure: Number; unit: participants
Arm/Group | Cidofovir
Number analyzed (Participants) | 32
participants | 14

6. Secondary Outcome: Identification of Abnormally Methylated Genes in Perianal Dysplasia
Description: Identification of abnormally methylated genes in perianal dysplasia
Time Frame: Baseline, after cycle 1, and 6 weeks after treatment discontinuation
Population: The lab analysis of genes was not performed
Arm/Group | Cidofovir
Number analyzed (Participants) | 0

7. Secondary Outcome: Distribution of Abnormally Methylated Genes Among HSIL, Low-grade Squamous Intraepithelial Lesions, and Normal Perianal Skin
Time Frame: Baseline, after cycle 1, and 6 weeks after treatment discontinuation
Population: The gene analysis was not done
Arm/Group | Cidofovir
Number analyzed (Participants) | 0

8. Secondary Outcome: Changes in Gene Expression in Perianal HSIL After Exposure to Cidofovir as Assessed by RNA Microarray Analysis
Time Frame: Baseline, after cycle 1, and 6 weeks after treatment discontinuation
Population: The gene expression analysis was not done
Arm/Group | Cidofovir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cidofovir
Serious Adverse Events (participants affected / at risk) | 3/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cidofovir (N=33)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dermatology/skin (Skin and subcutaneous tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cidofovir (N=33)
AST,SGOT Elevation (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Constitutional Symptoms (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dermatology/skin (Skin and subcutaneous tissue disorders) | 13 (21)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Fatigue (General disorders) | 3 (4)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Hemoglobinuria (Renal and urinary disorders) | 2 (4)
Hemorrhage, Anus (Blood and lymphatic system disorders) | 5 (7)
Hemorrhage, Rectum (Gastrointestinal disorders) | 2 (2)
Hemorrhage, other (Blood and lymphatic system disorders) | 4 (5)
Infection, other (Infections and infestations) | 3 (3)
Infection, lung (Infections and infestations) | 2 (2)
Infection, upper airway (Infections and infestations) | 2 (2)
Infection, vagina (Infections and infestations) | 2 (2)
Metabolic, other (Metabolism and nutrition disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 4 (11)
Neutropenia (Blood and lymphatic system disorders) | 3 (6)
Pain, other (General disorders) | 2 (3)
Pain, anus (Gastrointestinal disorders) | 9 (15)
Pain, back (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (General disorders) | 6 (7)
Pain, perineum (General disorders) | 14 (49)
Proteinuria (Renal and urinary disorders) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (21)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (3)
Ulceration (Skin and subcutaneous tissue disorders) | 12 (25)
Vomiting (Gastrointestinal disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Respiratory, thoracic, other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection, skin (Infections and infestations) | 6 (9)
Skin ulceration (Skin and subcutaneous tissue disorders) | 17 (30)
Upper respiratory infection (Infections and infestations) | 2 (2)
Vaginal infection (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No